CLINICAL TRIAL: NCT06656455
Title: Comparison of Two Anesthetic Protocols (Sevoflurane and Laryngeal Mask Airway Versus Propofol Infusion and Facemask) for Eye Examination Under Anesthesia in Children
Brief Title: Sevoflurane and Laryngeal Mask Airway Versus Propofol Infusion and Facemask for EUA in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Cynthia Karam, Principal Investigator, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANES.CK.01
Record Dates: First submitted 2024-10-21; First posted 2024-10-24 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia; Children, Only
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Active Comparator): Group S will be given propofol 2 mg/kg and fentanyl 1µg/kg intravenously and anesthesia will be maintained with sevoflurane via LMA
  Interventions: Drug: sevoflurane via LMA
- Group P (Experimental): Patients randomized to group P will be given propofol 1 mg/kg and fentanyl 1µg/kg intravenously and anesthesia will be maintained with a continuous infusion of propofol 200 µg/kg/min with oxygen 3 L/min via simple mask and oral airway if needed.
  Interventions: Drug: Propofol with oxygen via simple mask

INTERVENTIONS:
Drug: sevoflurane via LMA — In Group S, co-induction is used whereby the patient continues to receive 8% sevoflurane through the facemask followed after IV insertion by propofol 2mg/kg and fentanyl 1mic/kg administration. Thirty seconds afterwards, an age-appropriate LMA will be inserted. Sevoflurane is maintained initially at a concentration of 2%. The ventilation at first is assisted manually until the child starts breathing. If movement requires interruption of the exam, a bolus of propofol 1mg/kg is given and sevoflurane is increased by 1% until a maximal sevoflurane concentration of 4%. If apnea related to the depth of anesthesia occurs more than 10 sec or the saturation drops below 94%, sevoflurane will be turned off until the proper airway intervention is taken to achieve saturation above 95% and sevoflurane will be resumed at a concentration decreased by 1%.
  Arms: Group S
Drug: Propofol with oxygen via simple mask — In group P, the sevoflurane will be discontinued, and propofol 1 mg/kg and fentanyl 1µg/kg will be administered IV. Propofol pump is maintained initially at a rate of 200mic/kg/min. with oxygen at 3 liters/min via facemask.
  If movement requires interruption of the exam, a bolus of propofol 1mglkg is given and the infusion rate is increased by 20mic/kg/min up to a maximal rate of 350mic/kg/min. The total number of boluses needed will be recorded as the need for additional sedation. If apnea related to the depth of anesthesia occurs more than 10 sec or the saturation drops below 94%, the infusion pump will be stopped until the proper airway intervention is taken to achieve saturation above 95% with spontaneous breathing. Afterwards, the propofol pump will be resumed at a rate decreased by 20mic/kg/min.
  Arms: Group P

SUMMARY:
The goal of this clinical trial is to find out the optimal technique of anesthesia for eye examination in children. The main question it aims to answer is:

Is propofol infusion and simple oxygen facemask associated with earlier discharge from the operating room, and hence rapid turnover and greater efficiency compared to sevoflurane via LMA? Researchers will compare time to discharge from the operating room to see if eye examination for children less than 7 years using a propofol infusion pump based anesthesia and simple oxygen facemask results in a shorter discharge time from the operating room in comparison with sevoflurane via LMA.

Participants will will be assigned to receive general anesthesia by one of two treatment groups.

DETAILED DESCRIPTION:
Children younger than 5 years can be uncooperative during an examination and may render it impossible. The main objective of anesthesia for ophthalmic examination is to provide ideal conditions for optimal exam with a quick onset and offset of anesthesia as well as rapid recovery and early discharge. Two commonly used sedation techniques for young children are: sevoflurane via laryngeal mask airway (LMA) or propofol infused intravenously. Both have been shown to be safe and effective and allow rapid changes in anesthesia depth and minimal postoperative morbidity. However, their induction, emergence characteristics, and side effect profiles may differ. From previous studies, it is still not evident whether propofol infusion using oxygen facemask or sevoflurane administration via LMA is superior with respect to earlier discharge from operating room in children undergoing eye examination under anesthesia (EUA).

In the literature, there are no studies directly comparing those two different techniques for ophthalmic examination.

The aim of this study is to find out the optimal technique of anesthesia for eye examination in children resulting in earlier discharge from the operating room thus decreasing the turnover time between cases and providing optimal surgical conditions, without interfering with the well-being of the child or compromising the airway security.

In a prospective randomized study, a total sample of 60 children scheduled for eye examination under anesthesia (30 in each arm of the study) aged between 1-7 years with American Society of Anesthesiologists physical status 1 to 3 will be assigned to receive general anesthesia by one of two treatment groups. After induction with sevoflurane 8% in oxygen, patients randomized to group S will be given propofol 2 mg/kg and fentanyl 1µg/kg intravenously and anesthesia will be maintained with sevoflurane via LMA. Patients randomized to group P will be given propofol 1 mg/kg and fentanyl 1µg/kg intravenously and anesthesia will be maintained with a continuous infusion of propofol 200 µg/kg/min with oxygen 3 L/min via simple mask and oral airway if needed. In both groups sevoflurane concentration or propofol infusion will be titrated to keep optimal conditions. The primary outcome is time to discharge from the operating room. Secondary outcomes are surgical conditions, respiratory events, agitation and other side effects as well as recovery times. Normally distributed data will be summarized as mean ± SD and nonnormally distributed data will be summarized as median [interquartile range].

It is believed that propofol infusion and simple oxygen facemask will be associated with earlier discharge from the operating room, and hence rapid turnover and greater efficiency compared to sevoflurane via LMA. This study would have an impact on the current practice for pediatric ophthalmic EUA and may help find out the best technique that decreases the turnover time between cases resulting in higher operating time efficiency while providing optimal surgical conditions and patients' safety.

ELIGIBILITY:
Inclusion Criteria:

* Children presented to the Operating Room of the American University of Beirut Medical Center
* 1 to 6 years old
* With American Society of Anesthesiologists physical status 1-3
* Scheduled for ophthalmic EUA with or without laser/cryotherapy procedure

Exclusion Criteria:

* Children with full stomach or significant aspiration risk (including hiatal hernia)
* Children who are morbidly obese or have a current upper respiratory tract infection
* Children who have oropharyngeal pathology (e.g., radiotherapy for hypopharynx/larynx), tracheostomies, or a family history of malignant hyperthermia
* Children of parents who refuse to give consent
* Children having allergy to the anesthetics used
* Any surgical procedure expected to last for more than 60 minutes

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Time to discharge from the operating room | Time from the end of surgery to discharge from OR, assessed up to 40 minutes
  Time to discharge from the operating room in minutes

SECONDARY OUTCOMES:
Duration of anesthesia | From the start till the end of anesthesia, assessed up to 120 minutes
  Duration of anesthesia in minutes
Duration of surgical procedure | From the start of eye examination till the completion of the procedure, assessed up to 60 minutes
  Duration of surgical procedure in minutes
Ophthalmologist satisfaction score | During the procedure
  Ophthalmologist satisfaction score measured on likert scale (ranging from 1 till 5 with 1 representing the least degree of satisfaction and 5 the highest).
Apnea | During the procedure
  Apnea >10 seconds
Desaturation | During the procedure
  SPO2<94%
Laryngospasm | During the procedure
  Laryngospasm requiring treatment
Interruption | During the procedure
  Number of interruptions of EUA
Emergence agitation | Immediately after the procedure
  Emergence agitation on a four-point scale
Wake up time | Time from the end of anesthesia drug administration to spontaneous eye opening, assessed up to 180 minutes
  Wake up time in minutes
PACU stay duration | Time from arrival to PACU till achievement of an Aldrete score of 9, assessed up to 180 minutes
  PACU stay duration in minutes
Change in the airway management | Number of participants with change in airway management assessed by the data collector during the procedure
  Change in the airway management
Emesis | Number of participants who developed emesis, assessed by the data collector immediately after the procedure
  Emesis
Administration of pain medication | Number of participants who were administered pain medication, assessed by the data collector immediately after the procedure
  Administration of pain medication
Airway Obstruction | Number of participants who had an airway obstruction, assessed by the data collector during the procedure
  Airway Obstruction
Hypoventilation | Number of participants who developed hypoventilation, assessed by the data collector during the procedure
  Hypoventilation
Excess secretions | Number of participants who developed excess secretions, assessed by the data collector during the procedure
  Excess secretions
Induction time | Time from anesthesia start to surgery start, assessed up to 60 minutes
  Induction time in minutes
Nonoperative time | Time from anesthesia start to surgery start combined with the time to discharge from OR, assessed up to 60 minutes
  Nonoperative time in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Karam, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No